CLINICAL TRIAL: NCT00682942
Title: How to Predict Lung Recruitment at the Bedside in Patients Affected by Acute Lung Injury/Acute Respiratory Distress Syndrome (ALI/ARDS)
Status: Completed | Type: Observational
Sponsor: Policlinico Hospital (Other)
Responsible Party: Principal Investigator, Davide Chiumello, MD, Policlinico Hospital
Other Study IDs: 16500
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2011-12-01 (Estimated); Status verified 2011-11

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators aim to compare four different lung recruitment techniques (described in literature) to Computed tomography scan analysis.

DETAILED DESCRIPTION:
The investigators aim to compare four different lung recruitment techniques (described in literature) to Computed tomography scan analysis:

* stress index technique
* peep test
* recruitment technique used in the EXPRESS study
* recruitment technique used in the LOV study

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of acute lung injury/ acute respiratory distress syndrome
* Mechanical ventilation

Exclusion Criteria:

* Clinical diagnosis of chronic obstructive pulmonary disease
* Clinical diagnosis of pneumothorax
* Haemodynamic instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients affected by acute lung injury/acute respiratory distress syndrome who are mechanically ventilated
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2008-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Davide Chiumello, MD, Principal Investigator — Policlinico Hospital
Locations (1):
- Policlinico Hospital, Milan, Italy